CLINICAL TRIAL: NCT06468163
Title: Efficacy of Local Antibiotic Injection Via a Catheter for Treating Acute Periprosthetic Infections After Knee DAIR Surgery: A Prospective, Randomized Controlled Trial Study
Brief Title: Efficacy of Local Antibiotic Injection Via a Catheter for Treating Acute Periprosthetic Infections After Knee DAIR Surgery
Acronym: YES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Long Hua, Doctor, First Affiliated Hospital of Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HL240528-12
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Local Antibiotic Injection Catheter Acute Periprosthetic Infections Knee DAIR Randomized Controlled Trial
Keywords: Local Antibiotic Injection; Catheter; Acute Periprosthetic Infections; DAIR Surgery; Prospective; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter group (Experimental): Using catheter after knee DAIR surgery.
  Interventions: Device: Drug infusion into joint through catheter.
- None-catheter group (Active Comparator): Without using catheter after knee DAIR surgery.
  Interventions: Device: Drug infusion into joint through catheter.

INTERVENTIONS:
Device: Drug infusion into joint through catheter. — With or without using catheter after DAIR operation for drug infusion.

SUMMARY:
Prosthetic Joint Infection (PJI) is a severe complication following joint replacement surgery, imposing significant economic and health burdens on patients. For acute PJI, the DAIR (Debridement, Antibiotics, and Implant Retention) procedure is a necessary and effective treatment method, as it effectively clears the infection while preserving the prosthesis, thereby avoiding more complex surgical interventions. However, the practice of using drainage tubes postoperatively is controversial. Some studies suggest that drainage tubes may increase the risk of infection, while other literature indicates no statistically significant difference in infection risk associated with their use.In this context, Professor Li Cao's team at Xinjiang Medical University has improved the traditional DAIR procedure by incorporating long-term local antibiotic injections post-surgery, achieving positive results. Despite this, the specific method of antibiotic injection, particularly whether to use a drug infusion tube, remains under debate. The use of an infusion tube can reduce patient discomfort, shorten the local disinfection process, and theoretically decrease the time the incision is exposed to the external environment, potentially lowering the infection risk. However, the validity of these theoretical assumptions needs further confirmation through high-level scientific research. This study aims to evaluate whether there are differences in joint function recovery, changes in blood infection markers, and the incidence of postoperative complications between using and not using an infusion tube for local antibiotic injection after knee DAIR surgery. To assess the value of the infusion tube in local antibiotic injection post-knee DAIR surgery, a randomized controlled trial (RCT) will be conducted. Eligible patients will be randomly assigned to the infusion tube group (experimental group) or the non-infusion tube group (control group). The study will prospectively collect basic information, joint function scores, blood infection markers, and postoperative complication data from both groups, including patient age, gender, educational background, and postoperative blood test results. Ultimately, the RCT aims to demonstrate the therapeutic efficacy of the infusion tube method.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. Meet the diagnostic criteria for DAIR surgery of artificial knee joint;
3. Receiving knee DAIR surgery;
4. Voluntary and signed informed consent.

Exclusion Criteria:

1. Patients with chronic PJI infection undergoing total knee revision;
2. Patients with severe knee joint infection who cannot undergo artificial joint replacement;
3. Progressive renal insufficiency (stage 4 and above) or glomerular filtration rate less than 30ml/min;
4. periprosthesis infection after multiple joint replacement;
5. Active infection at the site of intravenous or joint injection;
6. long-term use of anticoagulants or antiplatelet drugs due to other diseases;
7. Have sepsis or positive blood culture within the last 30 days;
8. Radiotherapy and chemotherapy are required due to neoplastic diseases;
9. Receiving systemic glucocorticoid therapy (prednisone > 10mg/ day or equivalent hormone medication);
10. severe immunodeficiency diseases (such as stage 3 HIV, sickle cell anemia, splenectomy, etc.);
11. Have a history of drug abuse;
12. Treatment of bone marrow or other transplants with immunosuppressive drugs;
13. Pregnant, parturient and lactating women;
14. Participating in other clinical trials;
15. Researchers believe that other reasons are not appropriate for clinical trial participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection control rate | Two year after surgery
  Infection control rate
Time between infection recurrence | Two year after surgery
  Time between infection recurrence
Re-operation rate | Two year after surgery
  Re-operation rate

SECONDARY OUTCOMES:
X-ray | One day before surgery and two years after surgery
  X-ray
American Knee Society Score （AKS score） | One day before surgery and two years after surgery
  American Knee Society Score is used to evaluate the outcomes of knee replacement surgery. This scoring system consists of two main components: the knee score and the function score.
  Knee Score: This primarily assesses the condition of the knee joint itself, including pain, stability, and range of motion. The higher of the score, the better of the functional result.
Redness, Edema, Ecchymosis, Discharge, and Approximation score (REEDA score) | One day before surgery, three month after surgery
  The REEDA score is a clinical tool used to assess the healing of perineal wounds and other skin wounds, particularly after childbirth. REEDA stands for Redness, Edema, Ecchymosis, Discharge, and Approximation. Each of these five parameters is scored on a scale from 0 to 3, with higher scores indicating more severe symptoms. The total REEDA score can range from 0 to 15.
Visual Analog Scale score | One day before surgery and two years after surgery
  The VAS score, or Visual Analog Scale, is a tool commonly used to measure a person's level of pain. The VAS is a simple, subjective measure that consists of a straight line, typically 10 centimeters long, anchored by two endpoints. One end of the line represents "no pain" and the other end represents "worst pain imaginable." For example, if the VAS line is 10 cm long and the patient's mark is at 7 cm from the "no pain" end, their pain score would be 7 out of 10.
White blood cell count | One day before surgery and one day after surgery
  White blood cell count from blood
Erythrocyte sedimentation rate (ESR) | One day before surgery and one day after surgery
  It measures the rate at which red blood cells settle to the bottom of a test tube within one hour.
  Normal ranges:
  Male: 0 to 15 millimeters per hour (mm/hr) Female: 0 to 20 millimeters per hour (mm/hr)
C-reactive protein (CRP) | One day before surgery and one day after surgery
  C-reactive protein (CRP) is a protein produced by the liver that significantly increases in response to inflammation or infection. Normal range for CRP is less than 10 milligrams per liter (mg/L).
Synovial fluid white blood count | One day before surgery and one day after surgery
  Synovial fluid white blood count
Polymorphonuclear neutrophil percentage in synovial fluid (SF-PMN) | One day before surgery and one day after surgery
  Polymorphonuclear neutrophil percentage in synovial fluid refers to the proportion or percentage of polymorphonuclear neutrophils (PMN) present in the synovial fluid. This measurement is important in the assessment of joint health and inflammation, particularly in conditions such as arthritis and infections affecting the joints. Normal range: Less than 80%.
Alanine Aminotransferase (ALT) | One day before surgery and one day after surgery
  An enzyme found in the liver that helps convert proteins into energy. Elevated levels indicate liver damage. Normal range: 10 to 40 units per liter (U/L)
Aspartate Aminotransferase (AST) | One day before surgery and one day after surgery
  An enzyme found in the liver and other tissues. High levels can indicate liver damage but are less specific than ALT. Normal range: 10 to 40 units per liter (U/L)
Serum Creatinine | One day before surgery and one day after surgery
  Measures the level of creatinine in the blood. Elevated levels can indicate impaired kidney function. Normal range: 62 to 115 micromoles per liter (µmol/L).
Blood Urea Nitrogen （BUN） | One day before surgery and one day after surgery
  Measures the amount of nitrogen in the blood that comes from urea. Elevated BUN levels can indicate impaired kidney function. Normal range: 2.5 to 7.1 millimoles per liter (mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, M.D., Study Chair — The first affliated hospital, Xinjiang medical university

IPD SHARING:
Plan to Share IPD: Yes
Rawdata can be asked after paper published.
Supporting Information: Study Protocol
Time Frame: Rawdata can be asked after paper published.